CLINICAL TRIAL: NCT04527926
Title: Project STEPuP: A Prenatal Provider Education and Training Program to Improve Medication-assisted Treatment Use During Pregnancy and Maternal and Child Health Outcomes
Brief Title: STEPuP: Prenatal Provider Education and Training to Improve Medication-assisted Treatment Use During Pregnancy
Acronym: STEPuP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Krans, MD, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY19070128; 1R01DA049759-01 (NIH)
Record Dates: First submitted 2020-08-18; First posted 2020-08-27 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Opioid-use Disorder; Pregnancy Related
Keywords: Opioid-use Disorder; Medication-assisted Treatment; Pregnancy
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Postpartum Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STEPuP Intervention (Experimental): STEPuP interventions
  Interventions: Behavioral: STEPuP Intervention
- Usual Care (Active Comparator): Standard of Care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: STEPuP Intervention — Project STEPup has 4 components designed to address barriers to MAT and EBP adoption: 1) a "hub and spoke" remotely-supported provider education and training program, 2) addiction teleconsultation support, 3) case management and telepsychiatry support, and 4) a partnership with health system administrators and payers to address administrative and reimbursement related needs.
  Other Names: Project STEPuP(Substance abuse Treatment and Education during Pregnancy and Postpartum)
  Arms: STEPuP Intervention
Behavioral: Usual Care — Standard of Care
  Arms: Usual Care

SUMMARY:
This research will test the effectiveness of a prenatal provider education and training program designed to facilitate provider adoption of evidence-based practices for the treatment of OUD during pregnancy. Findings from this research will provide high quality evidence about how to increase evidence-based treatment for pregnant women with OUD and subsequent maternal-child health outcomes.

DETAILED DESCRIPTION:
The prevalence of opioid use disorder (OUD) during pregnancy has quadrupled over the past decade, as have maternal and neonatal morbidity and mortality related to substance use. Medication assisted treatment (MAT) use during pregnancy reduces adverse outcomes and is the recommended, evidence-based practice (EBP) for OUD treatment during pregnancy. Despite this, 40% of pregnant women with OUD do not receive MAT. Currently, there are no effective strategies to expand MAT access and availability for pregnant women, especially in rural, low-resource settings where maternal opioid use is disproportionately high. As an initial step to address this gap, the investigators engaged key stakeholders across a large health system in Pennsylvania to determine barriers and facilitators to expanding treatment services in high need, low-resource obstetric settings. The stakeholders identified a critical need for a women-centered, low resource, sustainable, provider-level intervention to facilitate the adoption of MAT in obstetric settings. Therefore, the investigators objective is to test the effectiveness of a prenatal provider education and training program designed to facilitate the adoption of EBP for OUD during pregnancy called Project STEPuP (Substance abuse Treatment and Education during pregnancy and Postpartum). Project STEPuP, grounded in preliminary and pilot work conducted by the research team, has 4 components designed to address barriers to MAT and EBP adoption: 1) a "hub and spoke," remotely supported provider education and training program, 2) addiction teleconsultation support, 3) case management and telepsychiatry support, and 4) a partnership with health system administrators and payers to address administrative and reimbursement related needs. To achieve this objective, the research team will conduct a cluster-randomized clinical trial across 12 obstetric sites in Pennsylvania and New York. Outcomes among 870 patients will be assessed during pregnancy, at delivery and through 1 year postpartum. The investigators central hypothesis is that Project STEPuP will facilitate EBP adoption, increase MAT utilization and improve health outcomes among pregnant and postpartum women with OUD and their children. Specifically, the investigators aim to: 1) Create organizational readiness to facilitate Project STEPuP implementation; 2) Assess the effect of Project STEPuP on provider adoption of EBP for OUD during pregnancy; and 3) Evaluate the effect of provider adoption of EBP on maternal and child health outcomes. The investigators research is significant by addressing the substantial knowledge gap of how to increase MAT use in pregnancy and innovative by examining the role that prenatal providers can play in expanding treatment access.

Study outcome measures refined in January 2024 to align with grant proposal and increase readability.

ELIGIBILITY:
Inclusion Criteria:

Providers:

1. provides prenatal care (i.e. obstetricians, nurse midwives, advanced practice providers) at obstetric sites,
2. provides care to pregnant women with OUD
3. English speaking

Patient:

Maternal and child outcome data will be collected from the Electronic Health Record (EHR) and individual patients will not be recruited to participate in the randomized controlled trial (RCT).

Inclusion criteria for a small subset of pregnant women will be recruited for a one-time qualitative interview (n=50):

1. meet The Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria for OUD
2. received care at participating sites while pregnant during the study time period and
3. speak English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient Medication-assisted treatment (MAT) utilization | up to 1 year post delivery
  As measured by total count of weeks in pregnancy with any Medications for Opioid Use Disorder (MOUD) either buprenorphine or methadone, use during pregnancy
Provider Provision of Buprenorphine | up to 1 year post delivery
  As measured by total number of patients within a prenatal practice with opioid use disorder that receive MOUD treatment (either buprenorphine or methadone)

SECONDARY OUTCOMES:
Hepatitis C Virus (HCV) Screening Rate | during pregnancy (up to 40 weeks)
  Number of participants screened for Hepatitis C Virus (HCV) as measured by related laboratory testing
Human Immunodeficiency Virus (HIV) Screening Rate | during pregnancy (up to 40 weeks)
  Number of participants screened for Human Immunodeficiency Virus (HIV) as measured by related laboratory testing
Mental Health Screening Rate | during pregnancy (up to 40 weeks)
  Number of participants who received a mental health screening test, Patient Health Questionaire-2 or Patient Health Questionaire-9 (PHQ-2 or PHQ-9)
Contraceptive Utilization Rate | delivery up to 1 year post delivery
  Number of participants utilizing postpartum contraceptive as measured by contraception prescription
Breastfeeding Rate | delivery up to 1 year post delivery
  Number of participants breastfeeding as measured by feeding records from infant charts (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Krans, MD, Principal Investigator — UPMC Magee-Womens Hospital; Marian Jarlenski, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No